CLINICAL TRIAL: NCT02517554
Title: A Randomized Study Of TeleGenetics Versus Usual Care To Increase Access To Cancer Genetic Services
Brief Title: A Study Of TeleGenetics Versus Usual Care To Increase Access To Cancer Genetic Services
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 09115
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Ovarian Cancer; Colorectal Cancer
Keywords: meet National Comprehensive Cancer Network® criteria for cancer genetic testing for breast, ovarian and colorectal cancers
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Remote cancer genetic services by videoconference
  Interventions: Behavioral: Penn genetic counselors provides counseling and test results disclosure by videoconferene to patient at community site
- Remote cancer genetic services by telephone
  Interventions: Behavioral: Penn genetic counselor provides counseling and test results disclosure by telephone to patient at community site
- Usual Care
  Interventions: Behavioral: Patient receives written information on how to find genetic services in their area

INTERVENTIONS:
Behavioral: Penn genetic counselors provides counseling and test results disclosure by videoconferene to patient at community site — Baseline and follow up survey
  Groups: Remote cancer genetic services by videoconference
Behavioral: Penn genetic counselor provides counseling and test results disclosure by telephone to patient at community site — Baseline and follow up surveys
  Groups: Remote cancer genetic services by telephone
Behavioral: Patient receives written information on how to find genetic services in their area — Baseline and follow up surveys
  Groups: Usual Care

SUMMARY:
The goal of this research is to evaluate the relative advantage of remote counseling over usual care in community health practices without access to genetic services. We will evaluate ability of remote telemedicine, referred to going forward as TeleGenetic services (phone or videoconferencing), to increase uptake of genetic testing and identification of genetic carriers compared to usual care. Secondly, we will evaluate the advantages of videoconferencing over telephone for delivery of remote genetic services and the short-term and longitudinal outcomes of TeleGenetic services in socio-demographically diverse patients in community practices.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants will include adult men and women (aged 18 and older) who can understand and communicate in English
2. meet National Comprehensive Cancer Network® criteria for cancer genetic testing for breast, ovarian or colorectal cancers
3. have insurance coverage for genetic testing.

Exclusion Criteria:

1. Under 18 years old - professional guidelines do not recommend genetic testing for cancer risk in minors.
2. Does not speak English.
3. Does not have insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Candidate for genetic testing for BRCA or colon cancer related genes
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-08; Primary Completion 2018-03 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Completion of Surveys | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bradbury, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (7):
- United States (7):
  - Union Hospital, Elkton, Maryland
  - Cape Regional Medical Center, Cape May Court House, New Jersey
  - Kennedy Health, Sewell, New Jersey
  - Shore Cancer Center, Somers Point, New Jersey
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Drexel Cancer Care at Hahnemann, Philadelphia, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania